CLINICAL TRIAL: NCT06213012
Title: Harnessing Neuroplasticity of Postural Sensorimotor Networks Using Non-Invasive Spinal Neuromodulation to Maximize Functional Recovery After Spinal Cord Injury
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Methodist Hospital Research Institute (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Principal Investigator, sayenko dimitry, Scientist, Associate Professor of Neurosurgery, The Methodist Hospital Research Institute
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PRO00037483; 5R01NS119587-02 (NIH)
Record Dates: First submitted 2023-10-26; First posted 2024-01-19 (Actual); Last update posted 2024-01-22 (Actual); Status verified 2024-01

CONDITIONS: Spinal Cord Injuries; Neuromodulation
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (3):
- Transcutaneous Spinal Stimulation (TSS) (Active Comparator): Spinal Stimulation delivered over the skin using a research stimulator with conventional surface electrodes during research visits.
  Interventions: Device: Transcutaneous Spinal cord Stimulation
- Sham (Sham Comparator): Sham Stimulation delivered over the skin using a research stimulator with conventional surface electrodes during research visits. Sham stimulation will be delivered using the intensity of stimulation set as during active sessions of ESS, but then gradually decreased down to zero in approximately 30 s. There will be 5-10 minute breaks interspersed between intervals of stimulation, and will vary according to the individual's tolerance and fatigue levels
  Interventions: Device: Transcutaneous Spinal cord Stimulation
- Epidural Spinal Stimulation (ESS) (Experimental): Stimulation delivered internally using an implanted device operated by an external control (only used during research visits).
  Interventions: Device: Epidural Spinal Stimulation (ESS)

INTERVENTIONS:
Device: Transcutaneous Spinal cord Stimulation — Delivered using a constant-current stimulator
  Arms: Sham; Transcutaneous Spinal Stimulation (TSS)
Device: Epidural Spinal Stimulation (ESS) — The device used for ESS, the CoverEdgeX 32 Surgical Lead system (Boston Scientific, USA), is a device approved by the FDA used in the treatment of severe pain and is approved for individuals to manage chronic pain when other treatments have not been effective.
  If you are in the ESS group, you will have surgery to have the stimulator placed and the stimulator will be removed at an office visit towards the end of the study.
  Arms: Epidural Spinal Stimulation (ESS)

SUMMARY:
It has been demonstrated that the human lumbosacral spinal cord can be neuromodulated with epidural (ESS) and transcutaneous (TSS) spinal cord stimulation to enable recovery of standing and volitional control of the lower limbs after complete motor paralysis due to spinal cord injury (SCI). The work proposed herein will examine and identify distinct electrophysiological mechanisms underlying transcutaneous spinal stimulation (TSS) and epidural spinal stimulation (ESS) to define how these approaches determine the ability to maintain self-assisted standing after SCI.

DETAILED DESCRIPTION:
Spinal circuitries below a paralyzing injury have a functional potential that far exceeds what has been thought possible. It has been demonstrated that task-specific motor therapy combined with epidural spinal cord stimulation (ESS) can promote improved motor function during postural, locomotor, and voluntary movement tasks, resulting in dramatic effects on the wellbeing of individuals with spinal cord injury (SCI). While these findings indicate a substantial promise for restoring mobility even after motor complete paralysis, chronic ESS is based on a high-cost implantable device, as well as an expensive and invasive surgical procedure. The investigators have developed a cost-effective alternative to ESS - non-invasive, transcutaneous electrical stimulation of the spinal cord (TSS). Preliminary works demonstrate that this neuromodulatory strategy provides sufficient specificity to selectively stimulate multisegmental dorsal nerve roots, enable stepping movements, and improve postural control during sitting and standing in individuals with motor complete SCI. The similarities between the effects of ESS and TSS are of critical importance in guiding more individually-specific neuromodulatory approaches to improve motor function and mobility after SCI, but have not been compared directly in the same subjects.

This study is focused on investigation the effects and mechanisms of each spinal neuromodulation strategy in regaining self-assisted standing. Not only is the recovery of balance control one of the most desired goals of people with paralysis, it provides the foundation necessary for regaining the ability to walk, and is critical to future therapies, involving robotic (e.g. exoskeleton) technologies. The objectives of this study are (1) to define the therapeutic potential of TSS during standing in individuals with motor complete SCI, and (2) to identify the neurophysiological and functional signatures of TSS and ESS. The central hypothesis is that each of the neuromodulatory strategies, when individually tailored, can result in significant motor recovery in individuals with chronic paralysis by reactivation and integration of networks that were clinically dormant prior to the intervention. The investigators predict that this proposal will have a high impact given that it encompasses multiple functional systems that contribute to the independence and quality of life in a broad population of individuals with SCI, and provides the first direct comparison of the invasive and non-invasive approaches. The investigators propose a progressive, mechanistic, and translational study to validate the effects of each approach, examine the neuroplastic capacity caused by activity-based training in the presence of TSS, and evaluate TSS and ESS stimulation paradigms as rehabilitative modalities after SCI.

ELIGIBILITY:
Inclusion Criteria:

* All participants must be able to provide a provision of a signed and dated informed consent form.

Stated willingness to comply with all study procedures and availability for the duration of the study.

* Male or female, aged 22-60 years old Able to provide paperwork from personal primary treating physician that proves stable medical condition with ability to tolerate at least 15 minutes upright
* Able to self-transfer from the wheelchair and demonstrate active range of motion of bilateral upper extremities in gravity dependent plane
* Able to passively range bilateral lower extremities within normal mobility parameters including: greater than 90 degrees of hip flexion and 165 degrees of hip extension; greater than 90 degrees of knee flexion and reach neutral knee extension of 180 degrees; neutral ankle position reaching a minimum of 90 degrees of dorsiflexion.
* Maintain current oral anti-spasticity regimen/dosage as approved by study physician with no change in regular use that may affect study outcomes.
* 1 to 6 years post spinal cord injury
* Non-progressive spinal cord injury
* Chronic motor complete SCI as defined by AIS A or B
* Neurological level of injury below T2 and above T10 (non-conus injury)
* Eligible for fMRI per safety questionnaire
* Women of childbearing potential must agree to the use of an effective means of avoiding pregnancy for the duration of the study.
* Able to commit to the full study

Exclusion Criteria:

* Currently involved in another rehabilitation training study
* Active pressure sores, unhealed bone fractures, peripheral neuropathies, or painful musculoskeletal dysfunction (including but not limited to contractures in the upper and lower extremities)
* Any ongoing medical condition which would preclude participant from regular physical activity (including but not limited to: cardiopulmonary disease, uncontrollable autonomic dysreflexia or orthostatic hypotension, active urinary tract infections, pregnant or nursing)
* Intrathecal baclofen pump therapy for spasticity
* Must not have received Botox injections to primary lower extremity and trunk musculature within the past 3 months, resulting in absence of muscle tone and precluding response to electrical stimulation therapy
* Current or history of neuromuscular conditions (including but not limited to: unhealed ligament of muscular tears in the upper or lower extremities, pain in weight bearing positions for upper and lower extremities).
* Clinically significant depression, psychiatric disorders, or ongoing drug abuse
* Any reason the PI or treating physician may deem as harmful to the participant to enroll or continue in the study
* Body Mass Index (BMI) over 30
* Pregnancy

Ages: 22 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-12-06 (Actual); Primary Completion 2027-08-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Assessment of force generation by lower limbs | Baseline 1(week 1), baseline 2(week 6), post interventions (week 11), and follow up (week 16)
  Neuromotor outcomes will be assessed during supine and upright standing, focusing on leg extension force output. Measurements will be taken under various conditions, including voluntary effort without spinal stimulation, and in the presence of Transcutaneous Spinal Stimulation (TSS), Epidural Spinal Stimulation (ESS), or Sham stimulation. The force output will be quantified in newtons (N). The magnitude of EMG signals will be quantified and expressed in millivolts (mV).

SECONDARY OUTCOMES:
Assessment of neurological status | Baseline 1(week 1), baseline 2(week 6), post interventions (week 11), and follow up (week 16)
  International Standards for Neurological Classification of SCI (ISNCSCI). The total motor score has a range of 0 to 100, with specific key muscles assessed on both sides of the body. The sensory scores also range from 0 to 112, evaluating light touch and pinprick sensation in different dermatomes.
Assessment of Independence | Baseline 1(week 1), baseline 2(week 6), post interventions (week 11), and follow up (week 16)
  Spinal Cord Independence Measure (SCIM). The SCIM involves assessing various neurological functions and assigning scores. The SCIM has a scale ranging from 0 to 100, with higher scores indicating greater independence in activities of daily living. The minimum score signifies complete dependence, while the maximum score reflects complete independence.

CONTACTS AND LOCATIONS:
Overall Officials: Dimitry Sayenko, MD, PhD, Principal Investigator — The Methodist Hospital Research Institute
Locations (1):
- Houston Methodist Hospital, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No